CLINICAL TRIAL: NCT02422056
Title: Acid Tranexamic Effectiveness in Reducing the Intraoperative Bleeding in Palatoplasty : Randomized Study
Brief Title: Acid Tranexamic Effectiveness in Reducing the Intraoperative Bleeding in Palatoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Guilherme Campelo Arantes, Guilherme Campelo Arantes MD, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1167-4683
Record Dates: First submitted 2015-03-31; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Cleft Palate; Hemorrhage
Keywords: Cleft Palate; Hemorrhage; Palatoplasty
MeSH Terms: conditions — Cleft Palate; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline infusion: Group receiving saline as placebo during the surgical procedure
  Interventions: Drug: Saline
- Intervention (Experimental): Tranexamic acid infusion: Group that received a Tranexamic acid bolus of 10mg / kg, followed by continuous infusion of 1 mg / kg / hr until the end of the procedure.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid bolus of 10 mg / kg at the beginning of palatoplasty, followed by infusion of 1 mg / kg / h until the end of the procedure
  Other Names: Transamin
  Arms: Intervention
Drug: Saline — Infusion of saline in the same rate used for the intervention group
  Other Names: Control
  Arms: Placebo

SUMMARY:
Randomized study evaluating the role of tranexamic acid in reducing intraoperative bleeding in palatoplasty.

DETAILED DESCRIPTION:
Double-blind randomized study comparing intraoperative bleeding in palatoplasty between patients who received tranexamic acid at a dose of 10mg / kg bolus followed by continuous infusion of 1 mg / kg / h until the end of the procedure and patients receiving placebo in similar arrangements.

Besides the impact on the volume of intraoperative bleeding the incidence of postoperative wound dehiscence in the first week and the incidence of oronasal fistulas after 1 month were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Palatoplasty indication in patients of any age with presence of congenital cleft palate (with or without associated cleft lip), in the study hospital

Exclusion Criteria:

* Preoperative hemoglobin lower than 10 mg / dl or platelet count less than 100,000 / mm3 ;
* Presence of coagulopathy caused by known coagulation cascade disorders or systemic diseases, or excessive bleeding history on previous occasions;
* History of bleeding disorders in first-degree relatives;
* Use of medications that may interfere with the coagulation cascade (platelet inhibitors or anticoagulants);
* Indication of secondary palatoplasty with the purpose of correction oro-nasal fistula;
* Known allergy to tranexamic acid.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding | during surgery
  Intraoperative bleeding volume defined as the sum of the volume of aspirated blood during the procedure and the volume of blood retained in the used gauze. The volume retained in the gauze was estimated by the difference between the dry weight and the weight after using them.

SECONDARY OUTCOMES:
Incidence of wound dehiscence | 5 days
  Presence of dehiscence of the surgical wound in partial or total plan of any extension, verified by clinical examination in the first postoperative return and photographic record. The existence of dehiscence was observed by the break in the suture line or extensive presence of fibrin in the wound bed (indicating open area at its base).
Oronasal fistulas | 1 month
  Presence of oronasal fistula type II, III or IV in pittsburgh classification verified on postoperative return at 1 month and photographic record.
incidence of significant bleeding complications | During hospital stay, an expected average of 2 days
  Incidence of bleeding requiring surgical intervention, blood transfusion or use of antifibrinolytic drugs in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme C Arantes, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP)